CLINICAL TRIAL: NCT03050658
Title: Skin Integrity After Newborns' First Bath And Development of Eczema and Allergy at 2 Years
Brief Title: Bathing Babies and Allergy
Acronym: BBA
Status: Completed | Type: Observational
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Ann Kellams, MD, Associate Professor, University of Virginia
Other Study IDs: 19587
Record Dates: First submitted 2017-02-06; First posted 2017-02-13 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Atopic Dermatitis; Allergy
MeSH Terms: conditions — Dermatitis, Atopic; Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — skin swabs
Oversight: Data Monitoring Committee: No

SUMMARY:
Atopic dermatitis (AD) is a chronic allergic skin disease with onset in early childhood and increasing prevalence in Westernized countries. Current well newborn guidelines for washing babies with soap were adopted by U.S. hospitals in the 1970s, before the rise in prevalence of allergic disease and AD (also called eczema). Increased transepidermal water-loss (TEWL) in newborn skin at 2 days of life was recently identified as a predictor of AD and allergy development by age 2 years. Risk for AD in babies was also linked to decreased skin colonization with certain skin microflora, such as staphylococcal organisms. Together, these data raise the question of whether newborn skincare guidelines have the potential to modify a baby's risk for allergy development. Our current practice of washing babies with soap may alter TEWL or other natural factors in skin that protect babies from development of AD and allergy. More knowledge is needed about the impact of infant skincare practices on allergy development.

The objective of this pilot study is to determine the impact of a baby's first bath on his/her transepidermal water loss (TEWL) and skin microflora. Study procedures will include collection of TEWL measurements and skin swabs for skin microflora analysis pre/post first bath in healthy term newborns at UVA. This data will serve as preliminary data for future studies.

DETAILED DESCRIPTION:
The UVA study team will perform all study-related procedures and will collect all data. Contact information and permission for the study team to contact the subject's family will be obtained at enrollment.

Pre-bath Procedures: Prior to the first bath, a study team member will:

1. Record health information about the subject.
2. Record the amount of vernix covering the subject's skin.
3. Measure skin TEWL (see TEWL below).
4. Procure skin swabs for microflora analysis (see Skin swabs below)

Post-bath Procedures: Following the subject's first bath, a study team member will repeat pre-bath procedures.

TEWL Procedure TEWL measurement will be performed using the Tewameter - a non-invasive, wand-like instrument that sits atop skin like a stethoscope and measures the water evaporating from the skin. TEWL is a validated non-invasive procedure for assessment of newborn skin integrity.

Skin Swabs Skin swabs, softer than Q-tips, will be wiped across the skin with soft pressure to allow transfer of the baby's skin microflora onto the swab for analysis of skin-colonizing microorganisms, according to established methods.

AD and allergy development by 2 years The medical charts of enrolled subjects will be reviewed at 24 months of life to determine the incidence of any physician-diagnosis of AD or allergic disease. Subjects who have no physician-diagnosis of AD or allergy in their medical record will be contacted according to the contact information they provided at enrollment. Investigators will get a medical release signed with informed consent so the study team can contact the PCP of the subject if they are not followed at UVA.

None of these procedures are part of routine care in newborns. All procedures are being done solely for research purposes and pose minimal risk to subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy term (>36 weeks GA) baby
* Born at UVA
* Admitted to the well newborn nursery
* Baby's mother is at least 18 years old and capable of providing informed consent

Exclusion Criteria:

* Babies born to cognitively-impaired mothers (unable to provide consent).
* Babies of prisoners.
* Babies of non-English speaking mothers (due to limited resources available for study conduct).
* Any other condition that in the opinion of the investigator would jeopardize the safety or rights of a participant or would render the participants unable to comply with the protocol.

Ages: 0 Hours to 72 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy term newborn babies admitted to the Well Newborn Service at the University of Virginia.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2017-02-07 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Change in skin transepidermal water loss (TEWL) | Within baby's first 72 hr of life, TEWL will be measured at baseline and then at 18 to 36 hours after their first bath in the hospital
  Change in TEWL, before (baseline) versus after baby's first bath, will be measured.

SECONDARY OUTCOMES:
Skin microorganisms | Within baby's first 72 hr of life, skin will be swabbed for microflora at baseline and then at 18 to 36 hours after their first bath in the hospital
  Skin will be swabbed for microflora analysis before and after baby's first bath
Number of participants with physician-diagnosis of atopic dermatitis and allergy | At 2 years of life, subjects will be assessed for any physician-diagnosis of atopic dermatitis (AD) or allergy during their first 24 months of life
  Prevalence of physician-diagnosed AD and allergy will be calculated among subjects at 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No